CLINICAL TRIAL: NCT06657768
Title: A Placebo-Controlled, Single- and Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, PK and PD of LY4006895 in Healthy Volunteers and Patients With Early Symptomatic AD
Brief Title: A Study of LY4006895 in Healthy Participants With Early Symptomatic Alzheimer's Disease (AD)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 27263; J5K-MC-OQAA (Other: Eli Lilly and Company)
Record Dates: First submitted 2024-10-23; First posted 2024-10-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease; Healthy
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- LY4006895 of Part A (SAD) (Experimental): Single-ascending doses of LY4006895 administered intravenously (IV)
  Interventions: Drug: LY4006895
- Placebo Part A (Placebo Comparator): Placebo administered IV
  Interventions: Drug: Placebo
- LY4006895 of Part B (MAD) (Experimental): Multiple-ascending doses of LY4006895 will be administered IV
  Interventions: Drug: LY4006895
- Placebo Part B (Placebo Comparator): Placebo administered IV
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY4006895 — Administered IV
  Arms: LY4006895 of Part A (SAD); LY4006895 of Part B (MAD)
Drug: Placebo — Administered IV
  Arms: Placebo Part A; Placebo Part B

SUMMARY:
The main purpose of this study is to evaluate the safety and tolerability of the study drug known as LY4006895. Part A will administer a single-ascending dose in healthy participants or Part B will administer multiple-ascending doses in participants with early symptomatic Alzheimer's Disease (AD).

Blood tests will be performed to check how much LY4006895 gets into the bloodstream and how long it takes the body to eliminate it.

This is a 2-part study and will last approximately 29 weeks for Part A and 61 weeks for Part B, including a screening period for each part.

ELIGIBILITY:
Inclusion Criteria for Part A and Part B:

* Are overtly healthy as determined by medical evaluation. Rescreening is not allowed in this study
* Have a body mass index (BMI) within the range 18 to 40 kilogram per square meter (kg/m²)

For Part A:

* Have early symptomatic AD, as defined by:

  * Gradual and progressive change in memory function for at least 6 months, as reported by the participant or informant
  * A Mini-Mental State Exam (MMSE) score of 18 to 30 at screening
  * A Clinical Dementia Rating (CDR) global score of 0.5 to 1.0 (inclusive), with a memory box score greater than or equal to 0.5 at screening

For Part B:

* Have up to 2 reliable study partners who are in frequent contact with the participant (defined as at least 10 hours per week), one of whom at any one occasion: will accompany the participant to the study visits, will be available by telephone at designated times, and will provide a separate written informed consent to participate

Exclusion Criteria for Part A and Part B:

* Current serious or unstable illnesses including cardiovascular, hepatic, renal, gastroenterological, respiratory, endocrinologic, neurologic (MAD: other than AD), psychiatric, immunologic, or hematologic disease and other conditions that, in the investigator's opinion, could interfere with the participant's ability to complete the study; or has a life expectancy of less than 24 months
* Have screening hemoglobin (Hb) less than 12 grams per deciliter (g/dL) or evidence of iron-deficiency (ferritin less than 30 nanograms per milliliter (ng/mL), or presence/history of hemoglobinopathy
* Are, in the judgment of the investigator, actively suicidal and therefore deemed to be at significant risk for suicide
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening that cannot be explained by regular concomitant medications
* Have previous exposure to any anti-tau therapy
* Are pregnant or intend to become pregnant or to breastfeed during the study

For Part B:

* Have a current exposure to an amyloid targeted therapy. Prior exposure to amyloid targeted therapies greater than 1 year from the last dose may be permitted at the discretion of the investigator and in consultation with the sponsor. A listing of amyloid targeted therapies will be provided
* Have a sensitivity to florataucipir 18F
* Have contraindication to magnetic resonance imaging (MRI) including claustrophobia or the presence of contraindicated metal (ferrogmagnetic) implants/cardiac pacemaker

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with One or More Treatment Emergent Adverse Events (TEAEs), Serious Adverse Event(s) (SAEs), and Discontinuations due to Adverse Event(s) (AEs) Considered by the Investigator to be Related to Study Drug Administration | Baseline to Study Completion (Up to 61 Weeks)
  A summary of TEAEs, SAEs, and AEs regardless of causality, will be reported in the Reported Adverse Events module

SECONDARY OUTCOMES:
PK: Maximum Concentration (Cmax) of LY4006895 | Baseline to Study Completion (Up to 61 Weeks)
  PK: Cmax of LY4006895
PK: Area Under the Concentration Versus Time Curve (AUC) of LY4006895 | Baseline to Study Completion (Up to 61 Weeks)
  PK: AUC of LY4006895

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- United States (7):
  - Collaborative Neuroscience Network - CNS, Los Alamitos, California
  - K2 Medical Research - The Villages, Lady Lake, Florida
  - K2 Medical Research, Maitland, Florida
  - Atlanta Center of Medical Research, Atlanta, Georgia
  - CenExel iResearch, LLC (CenExel iRA), Decatur, Georgia
  - CenExel-HRI, Marlton, New Jersey
  - Duke Early Phase Research Unit, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No